CLINICAL TRIAL: NCT00175162
Title: A Comparison of Fixation Method in Total Knee Arthroplasty - Low Viscosity Versus High Viscosity Bone Cement. A Prospective Randomized Migration- and Bone Density Study on Primary Cemented Knee Implants.
Brief Title: A Comparison of Fixation Method in Total Knee Arthroplasty - Low Viscosity Versus High Viscosity Bone Cement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No financing possible
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20030249
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2010-10

CONDITIONS: Osteoarthritis
Keywords: RSA; DEXA; Genoarthrosis; Knee Arthroplasty; Micromotion of polyethylene liner; Cement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopal G bone cement (Active Comparator)
  Interventions: Device: Osteopal G vs. Refobacin-Palacos R bone cement
- Refobacin-Palacos R bone cement (Active Comparator)
  Interventions: Device: Osteopal G vs. Refobacin-Palacos R bone cement

INTERVENTIONS:
Device: Osteopal G vs. Refobacin-Palacos R bone cement — Bone cement
  Other Names: Osteopal G bone cement; refobacin-palacos R bone cement

SUMMARY:
The purpose of this study is to compare the early migration and periprosthetic bone changes of two total knee arthroplasties fixated with two different type bone cement.

DETAILED DESCRIPTION:
Around 4% of total knee arthroplasties (TKA) are revised 15 years after the primary operation, most due to loosening of the implant. About 70 % TKA are fixed with bone cement and in general the results after total knee arthroplasty are excellent and with the existing technique about 95% well functioning prostheses can be expected 10 years post surgery. The most serious late complication to surgery is aseptic loosening of the implants; and this remains one of the main courses of failure of both uncemented and cemented total knee implants.

Implant design, method of fixation, the quality of bone cement, surgerytechnique and the bone mass density are some of the factors that have a large influence on implant stability. Fixation of the tibia baseplates in total knee arthroplasty can be obtained by different type bone cement.

In this project we are using a modular tibia component with a central wedge-shaped stem. Upon randomization at surgery the implant is consolidated in the bone with either low-viscosity or high-viscosity bone cement.

The purpose of this study is to compare the early migration of a total knee implant fixated with two different bone cements using RSA (radio stereophotogrammetric analysis) for evaluation. Furthermore, we will make research into the periprosthetic bone and its changes post surgery using DEXA. Finally, the extend of the expected micromovements between the polyethylen liner and the metal backing of the titanium plateau will be compared and taken into account with the results.

Several factors can influence the long-term survival of cemented TKA. Bone-sclerosing at the tibia condyles may induce a problem with cement penetration into the cancellous bone. Furthermore, blood-contamination in the cancellous bone may reduce the shear-strength at the bone-cement site by 50%. A solid cement-implant interface limits the amount of debris in the interface bringing down the risk of radiolucent lines and osteolysis. The tibial implant used in this study is designed with a rim under the plateau to support the cement layer on the tibial condyles at the time of fixation. The implant has a stem making it more resistant to shearing forces. In this study we primarily consider the bone cement viscosity on the outcome. Both types are used in hip-arthroplasties with good results.

To evaluate both the implant-bone micromotions and the polyethylen-implant micromovements metal markers have been placed on the tibial implants pre-operatively. They will also be inserted into the tibial bone and into the tibial polyethylen intra-operatively allowing us to evaluate stereo x-rays by a photogrammetric computer analyses called RSA at the Orthopaedic Center, Aarhus University Hospital. Follow-up stereo x-rays will be scheduled for 1 week, 3 months, 6 month, 1 years and 2 years post-surgery. Periprostetic bone density will be evaluated at 1 week, 1 year and 2 years upon inclusion at the Orthopaedic Center, Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one- or double-sided primary knee arthrosis.
* Patients with a sufficient bone quality for implantation of knee prosthesis.
* Informed and written patient consent.

Exclusion Criteria:

* Patients with neuromuscular or vascular diseases in the affected leg.
* Patients who peroperatively are estimated unsuitable for knee arthroplasty e.g. due to bone cysts or dilution of the bone mass.
* Patients who use non-steroid anti-inflammatory drugs (NSAID) and cannot refrain from taking them postoperatively (this includes COX-2-inhibitors).
* Patients with osteoporosis estimated from the preoperative x-ray or former diagnosis of osteoporo-sis.
* Patients with knee arthrosis following fracture sequelae.
* Women, who are pregnant or are at risk of getting pregnant throughout the 2 year follow-up.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2010-12

PRIMARY OUTCOMES:
Tibial prosthesis part migration evaluated by RSA. | 2011

SECONDARY OUTCOMES:
Micromotion of the modular polyethylen liner in both type prostheses evaluated by RSA estimating the role of wear. | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD, Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Tage-Hansens Gade 2, 8000 Aarhus C, Denmark.
Locations (1):
- Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark